CLINICAL TRIAL: NCT00062842
Title: Pediatric Phase I and Pharmacokinetic Study of Irinotecan
Brief Title: Study of Irinotecan on a Weekly Schedule in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Susan Blaney, Professor, Pediatrics-Hema & Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H6957
Record Dates: First submitted 2003-06-17; First posted 2003-06-18 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Irinotecan; irinotecan sucrosofate

ARMS (1):
- Irinotecan weekly (Experimental): Irinotecan was administered over 90 min weekly 4x, every 6 weeks.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan
  Other Names: Onivyde,

SUMMARY:
The medicine being offered in this study is called Irinotecan. Irinotecan has been effective against many animal cancers. It has been given to both adults and children. We are now attempting to determine how much of the drug can be given to children when Irinotecan is given weekly for four weeks in a row every 6 weeks and the toxicities (bad side effects) that occur when irinotecan is administered on this schedule.

The purposes of this study are to:

1. To determine the highest dose of Irinotecan that can safely be given to children whose cancer no longer responds to standard treatment.
2. To determine the toxicities of Irinotecan.
3. To determine what studies (laboratory or x-rays) need to be done to evaluate the toxicities of this drug.
4. To determine if irinotecan is beneficial to the patient.
5. To understand how the drug Irinotecan works in the body.

DETAILED DESCRIPTION:
Irinotecan will be given intravenously (into the vein) over 90 minutes for four weeks in a row. This cycle may be repeated in six weeks as long as the cancer is not getting worse and there are no serious side effects.

After one cycle patients will be evaluated to decide if the treatments should continue. If the disease is no worse or better additional courses may be given. If treatment continues, evaluations will be done after the second cycle and then every 2 cycles.

If patients choose to participate in this study we would request that they remain in the study for one full cycle. During the first cycle of treatment we would like to draw special blood samples to help us learn how much drug is in the blood. These special studies are called pharmacokinetics. On the first day the drug is given, fourteen blood samples will be drawn. Each blood sample will be about 1/2 teaspoon, for a total of about 3 tablespoons. These samples will only be drawn during the first cycle of therapy. The total amount of blood drawn will be less than 5% of the total blood volume, an amount safe even for small children.

Examinations and other blood tests will be done twice a week initially, then weekly to look for side effects of the drug. Patients will have an additional one teaspoon of blood drawn at each of these visits.

ELIGIBILITY:
Stratum 1 Eligibility Criteria

* Must be ≥ 1 and ≤ 21 years of age.
* Must have histologically or cytologically documented diagnosis of solid tumor refractory to conventional therapeutic modalities or for which no effective therapy is known. Patients with brain tumors will be eligible for this study. For patients with brain stem gliomas the requirement for histologic verification may be waived.
* Must have evaluable disease. Evidence of measurable disease on radiographic studies is not required for entry onto the protocol.
* Karnofsky ≥ 50% for patients > 10 years of age and or Lansky ≥ 50% for children ≤ 10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
* Patients must have a life expectancy of at least 8 weeks.
* Patients must have recovered from the acute toxic effects of all prior therapy.
* Myelosuppressive chemotherapy: Must not have received within 3 weeks of entry onto this study (six weeks if prior nitrosourea)
* XRT: ≥ 6 months must have elapsed if prior craniospinal XRT or if ≥ 50% radiation of pelvis; ≥ 6 wks must have elapsed if other substantial BM radiation
* Autologous BMT without TBI: ≥ 6 mos must have elapsed (if applicable). Does not include prior treatment with high dose chemotherapy followed by stem cell rescue.
* Growth factor(s): Must not have received within 1 week of entry onto this study
* Patients with brain tumors who are receiving dexamethasone must be on a stable or decreasing dose for at least 2 weeks prior to study entry.
* Must have adequate bone marrow function (peripheral ANC ≥ 1,500/mm3, platelet count ≥ 100,000/mm3; hemoglobin ≥ 8.0 g/dl.)
* Must have adequate renal function (normal creatinine for age or GFR ≥ 70 ml/min/1.73m2) and hepatic function (bilirubin < 1.5 mg/dl; SGPT < 5x normal).

Stratum 1 Exclusion Criteria:

* Patients who have previously received irinotecan.
* Patients who are pregnant or lactating. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Patients who have an uncontrolled infection.
* Patients who are receiving any other cancer chemotherapy or any other investigational agents.
* Patients who have had a BMT which included TBI or an allogeneic BMT.
* Patients with bone marrow involvement.
* Patients who are receiving anticonvulsants as outlined in stratum 3.

Stratum 2:

* Stratum 1 must be closed. All patients who fulfill the Eligibility Criteria for Stratum 1and the Exclusion Criteria plus the following exclusions:
* Patients who have received more than two prior multi-agent chemotherapy regimens.
* Patients who have had prior central axis radiation.
* Patients who have had bone marrow transplantation (with or without TBI).
* Patients who have had pelvic, and/or total abdominal radiation.

Stratum 3:

* Patients receiving enzyme inducing anticonvulsants ( phenytoin, phenobarbital, carbamazepine, etc.) are eligible for this study if they meet the eligibility and exclusion criteria for the corresponding open stratum (Stratum 1 or 2).
* Patients must be on a stable dose of their anticonvulsant medication for a minimum of two weeks prior to study entry.
* Patients who are taking valproic acid must also be receiving another enzyme inducing anticonvulsant drug in order to be eligible for the study.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 1998-09-09 (Actual); Primary Completion 2005-05 (Actual); Study Completion 2006-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States